CLINICAL TRIAL: NCT05375006
Title: Tropism and Pathogenesis of Influenza Virus and Coronavirus in Human Brain Explant Culture
Acronym: COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Owen Ho KO, Assistant Professor, Chinese University of Hong Kong
Other Study IDs: 2022.120
Record Dates: First submitted 2022-05-12; First posted 2022-05-16 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Influenza Virus; Coronavirus
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Brain Tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background:

Influenza and coronavirus have been repeatedly causing pandemic recently. Like the Influenza A/H7N9 virus has caused five epidemics in China since its first detection in East China in 2013. In 2017, the previously low pathogenic avian influenza (LPAI) H7N9 virus underwent mutation in its haemagglutinin to give to a highly pathogenic avian influenza (HPAI) virus causing 32 human cases and potentially poses a threat to animal and human health. More recently, the SARS-CoV-2 pandemic has been heavily affecting the world. Therefore an effective risk assessment platform is urgently required for better pandemic preparation.

Hypothesis:

The tissue tropism and pathogenesis of a newly emerged infectious viruses, like the highlypathogenic influenza, like H7N9 and coronavirus, like SARS-CoV-2 would be different from that of their low pathogenic subtype and it would infect and replicate the human respiratory system more efficiently.

Because of its resistance to oseltamivir for influenza and no effective antiviral for coronavirus, investigators therefore propose to set up an novel and effective risk assessment platform for emerging infectious viruses.

Experimental Design:

The tissue tropism and viral replication kinetics of a HPAI and LP influenza and coronavirus will be determined in ex vivo cultures of human brain and compared with their LP subtype. The replication competence and innate immune responses of influenza and coronavirus will be studied and compared with other LP virus in in vitro cultures of human brain cells and human microvascular endothelial cells (HMVEC) both isolated from human brain tissues.

Expected outcomes:

HPAI influenza and coronavirus particularly SARS-CoV-2 will infect and replicate the human brain tissues and cells more efficiently than their LP subtype. Besides, HPAI influenza and SARS-CoV-2 will induce dysregulated host innate immune response than the LP subtype.

DETAILED DESCRIPTION:
In this study, 80 subjects who will undergoing elective or emergency craniotomies for intrinsic brain lesions at Prince of Wales Hospital, will be recruited.

This is a prospective and qualitative study. There is no randomization in the study procedure nor therapeutic invention for study subjects. No investigational product is involved.

Brain tissues that are normal discarded during the operation from patients who undergo elective or emergency craniotomies for intrinsic brain lesions will be collected for this study.

A consent for operation and agreement to use of removed tissue for scientific research will be obtained prior to the procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Age: > 1 year old and < 70 years old
2. Undergo elective or emergency craniotomies for intrinsic brain lesions

Exclusion Criteria:

a. Samples containing infected material

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will recruit participants who will undergoing elective or emergency craniotomies for intrinsic brain lesions at Prince of Wales Hospital
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-05-26 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Replication kinetics of influenza virus using ex vivo cultures of human brain | baseline
  Tissue fragments will be infected with 106 TCID50/mL for 1h at 37°C and then washed with 3 ml of warm PBS for three times to remove unbound virus. To determine productive viral replication from the infected biopsy specimens, supernatants of the infected cultures will be collected at 1, 24, 48 and 72hpi and virus titers will be determined by TCID50 assay. Explant cultures will be fixed in 10% formalin at 24 and 72hpi and immunohistochemistry staining (IHC) against HB65 antibody (European Veterinary Laboratories), SARS-CoV or SARS-CoV-2 viral antibody will be performed for the detection of virus-infected cells.
replication efficiency and innate immune responses of influenza virus | baseline
  Cells will be infected with viruses at either MOI of 0.01 or 2 for 1h. After 1h virus adsorption, viruses will be aspirated and cells will be washed with PBS for three times, then medium will be replenished. For cells infected at MOI of 0.01, cell culture supernatant will be harvested at 1, 24, 48 and 72hpi and viral titers will be determined by TCID50 assay.
Replication kinetics of coronavirus using ex vivo cultures of human brain | Baseline
  Tissue fragments will be infected with 106 TCID50/mL for 1h at 37°C and then washed with 3 ml of warm PBS for three times to remove unbound virus. To determine productive viral replication from the infected biopsy specimens, supernatants of the infected cultures will be collected at 1, 24, 48 and 72hpi and virus titers will be determined by TCID50 assay. Explant cultures will be fixed in 10% formalin at 24 and 72hpi and immunohistochemistry staining (IHC) against HB65 antibody (European Veterinary Laboratories), SARS-CoV or SARS-CoV-2 viral antibody will be performed for the detection of virus-infected cells.
replication efficiency and innate immune responses coronavirus | Baseline
  Cells will be infected with viruses at either MOI of 0.01 or 2 for 1h. After 1h virus adsorption, viruses will be aspirated and cells will be washed with PBS for three times, then medium will be replenished. For cells infected at MOI of 0.01, cell culture supernatant will be harvested at 1, 24, 48 and 72hpi and viral titers will be determined by TCID50 assay.

CONTACTS AND LOCATIONS:
Overall Officials: Owen Ho Ko, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, NT, Hong Kong

IPD SHARING:
Plan to Share IPD: No